CLINICAL TRIAL: NCT07048405
Title: Investigating the Cellular Heterogeneity of Human Brown Adipose Tissue and Its (Patho)Physiological Regulation
Brief Title: Intermittent Cold Exposure and Brown Adipose Tissue Hyperplasia
Acronym: ICEBATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 350117; 24/SS/0094 (Other: Health Research Authority (HRA))
Record Dates: First submitted 2025-05-06; First posted 2025-07-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Brown Adipose Tissue; Cold Exposure; 18F-FDG PET/CT
Keywords: Brown Adipose Tissue; Cold Exposure; 18F-FDG PET/CT
MeSH Terms: interventions — Cool-Down Exercise; Biopsy; Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy normal weight subjects (Experimental)
  Interventions: Other: Cooling; Procedure: Biopsies; Radiation: Injection of 18F-FDG; Other: Indirect calorimetry; Other: Electromyogram; Other: Core and skin temperature monitoring

INTERVENTIONS:
Other: Cooling — Participants will undergo cold exposure during the baseline and final visits (2.5 hours each visit), as well as throughout the 10-day cold acclimation period (2 hours per day). This will be achieved using water-perfused blankets set to individualized temperatures, selected to elicit comparable physiological responses across participants.
Procedure: Biopsies — Under local anesthesia, biopsies will be obtained from the following sites:
  * Brown adipose tissue from the supraclavicular (collarbone) region, guided by computed tomography (CT).
  * White adipose tissue from the abdominal (periumbilical) area.
  * Skeletal muscle from the outer thigh, specifically the vastus lateralis.
  These biopsies will be performed both before and after the 10-day cold acclimation protocol.
  Other Names: brown adipose tissue biopsy; white adipose tissue biopsy; skeletal muscle biopsy
Radiation: Injection of 18F-FDG — Intravenous injection of 18F-FDG will be performed after 2 hours of cold exposure. This will be followed by a 30min dynamic total PET/CT scan while cold exposed using water-perfused blankets. These procedures will take place before and after the 10 day-cold acclimation protocol.
Other: Indirect calorimetry — Participants will rest quietly while oxygen consumption and carbon dioxide production are continuously recorded using a indirect calorimeter. These data will be used to calculate energy expenditure and respiratory exchange ratio. This procedure will take place before and after the 10 day-cold acclimation protocol.
Other: Electromyogram — Skin surface electrodes will be placed on major skeletal muscles to measure shivering and muscle activity during both warm and cold conditions. This procedure will take place before and after the 10 day-cold acclimation protocol.
Other: Core and skin temperature monitoring — Participants will ingest an electronic capsule that wirelessly and continuously monitors core body temperature. This procedure will be conducted before and after the 10-day cold acclimation protocol.
  Additionally, wireless temperature sensors will placed at multiple standardized sites on the body to measure skin temperature. This procedure will be performed before, during, and after the 10-day cold acclimation protocol.

SUMMARY:
This clinical trial explores how repeated short-term cold exposure impacts the molecular and physiological function of brown adipose tissue (BAT), a thermogenic organ associated with improved cardiometabolic health. While intermittent cold exposure has been shown to increase BAT activity and mass, as measured by fluorodeoxyglucose (18F-FDG) uptake on positron emission tomography/computed tomography (PET/CT) scans, the molecular adaptations within BAT and other thermogenic tissues including skeletal muscle and white adipose tissue (WAT) remain poorly understood.

Healthy adults aged 18 to 40 years (6 males and 6 females) will participate in a 10-day cold acclimation protocol (2 hours per day using water-perfused cooling blankets). The primary objective is to determine how cold exposure alters cellular heterogeneity and gene expression in BAT, WAT, and skeletal muscle.

Participants will undergo baseline assessments, including measurements of energy expenditure, core and skin temperature, muscle activity, and blood sampling, each performed in both warm and cold conditions. These assessments will be followed by dynamic total-body PET/CT imaging during cold exposure and tissue biopsies from BAT, subcutaneous WAT, and skeletal muscle. These procedures will be repeated after the cold acclimation protocol to evaluate physiological and molecular changes. Additional outcomes include changes in energy expenditure, cold tolerance, and immune cell responses induced by cold exposure.

DETAILED DESCRIPTION:
Twelve healthy adults aged 18-40 years old (6 female, 6 male) will:

* Attend baseline visits in both warm and cold conditions for blood sampling, measurement of energy expenditure, skin and core temperature, muscle activity. This will be followed by dynamic total-body 18F-FDG PET/CT scan during cold exposure.
* Undergo biopsies of BAT (supraclavicular), skeletal muscle (vastus lateralis), and subcutaneous WAT (periumbilical) under local anesthesia.
* Complete 10 consecutive days of cold acclimation (2 hours per day) using water-perfused cooling blankets.
* Return for follow-up assessments, including repeat blood sampling, energy expenditure, temperature measurements, PET/CT imaging, and tissue biopsies to evaluate post-acclimation changes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years
* Body mass index 18.5-25 kg/m2
* Weight change of less than 5% in the past 6 months
* No acute or chronic medical conditions
* On no regular medications (other than contraceptives in female participants)
* No claustrophobia
* Alcohol intake ≤14 units/ week
* Screening blood tests within acceptable limits (of no clinical significance)
* Not currently pregnant, lactating or breastfeeding (female participants only)
* Ability to provide informed consent.

Exclusion Criteria:

* Not meeting inclusion criteria
* Contra-indication to PET/CT scan
* Allergy to local anaesthetic

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tissue transcriptional changes derived from cold exposure | 1 year
  We will be analysing and comparing gene expression from nuclei extracted from BAT, WAT and skeletal muscle before and after cold the 10-day cold acclimation protocol.

SECONDARY OUTCOMES:
Changes in brown adipose tissue activity/mass before and after cold acclimation protocol | year after
  BAT activity/mass will be measured using the glucose analogue 18-FDG radiotracer combine with PET/CT.
Energy expenditure | year after
  Energy expenditure measured with indirect calorimetry before and after cold acclimation protocol to evaluated any changes in response to intermittent cold exposure.
Skin and core temperature | year after
  Measurement of skin and core temperature before and after the cold acclimation protocol
Immune cell levels | year after
  Analyse the percentage of immune cell populations before and after cold acclimation

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No